CLINICAL TRIAL: NCT03541187
Title: Cockroach Immunotherapy in Children and Adolescents
Acronym: CRITICAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ICAC-28; UM1AI114271 (NIH); NIAID CRMS ID#: 38517 (Other: DAIT NIAID)
Record Dates: First submitted 2018-05-07; First posted 2018-05-30 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Persistent Asthma
Keywords: cockroach; immunotherapy; inner city asthma; subcutaneous immunotherapy (SCIT); Nasal Allergen Challenge (NAC)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G. cockroach allergenic extract (Experimental): Subcutaneous immunotherapy (SCIT): German cockroach allergenic extract. 40 participants 8 to 14 years of age will be randomized to this treatment arm.
  -Up to 2 doses of the assigned SCIT treatment will be given weekly during dose escalation, separated by a minimum of 2 days. After maintenance dose is achieved, participants will receive three maintenance level-doses spaced approximately 2 weeks apart, followed by maintenance injections every 4 weeks for the remainder of the treatment period. The treatment is for a period of 12 months.
  Interventions: Biological: German cockroach allergenic extract
- Placebo (Placebo Comparator): Subcutaneous immunotherapy (SCIT): Placebo for German cockroach allergenic extract. 40 participants 8 to 14 years of age will be randomized to this treatment arm.
  -Up to 2 doses of the assigned SCIT treatment will be given weekly during dose escalation, separated by a minimum of 2 days. Once the maintenance dose is achieved, participants will receive three maintenance level-doses spaced approximately 2 weeks apart, followed by maintenance injections every 4 weeks for the remainder of the treatment period. The treatment is for a period of 12 months.
  Interventions: Biological: Placebo for German cockroach allergenic extract

INTERVENTIONS:
Biological: German cockroach allergenic extract — Active ingredient: a non-standardized allergen derived from the extraction and purification of proteins from German cockroach (Blattella germanica). Non-standardized glycerinated German cockroach allergenic extract is approved in the United States for diagnostic skin testing and immunotherapy by subcutaneous injection (U.S. License 467).
  Other Names: Blattella germanica allergenic extract
  Arms: G. cockroach allergenic extract
Biological: Placebo for German cockroach allergenic extract — Commercially- labeled licensed product, sterile diluent for allergenic extract (50% glycerinated), sodium bicarbonate (0.091%) sodium chloride (0.166%).
  Other Names: Placebo for Blattella germanica allergenic extract
  Arms: Placebo

SUMMARY:
Scientific evidence has shown that, over the past two decades, the combination of cockroach allergy and cockroach exposure is one of the most important factors contributing to the dramatic increase in asthma morbidity seen in inner city children with asthma. Therefore, a major goal of the Inner City Asthma Consortium (ICAC) is to evaluate the efficacy of cockroach immunotherapy in inner city asthma.

The primary objective of the study is to determine if the response to nasal allergen challenge (NAC) will be changed with treatment with cockroach subcutaneous immunotherapy (SCIT) treatment.

DETAILED DESCRIPTION:
This is a 1:1 randomized, double-masked (blind), placebo-controlled, multicenter trial with 2 treatment arms:

* German Cockroach Subcutaneous Immunotherapy (SCIT) + guideline-based standard asthma care, OR
* Placebo (for German Cockroach Subcutaneous Immunotherapy [SCIT]) + guideline-based standard asthma care

Eighty participants 8 to 17 years of age who are sensitized to cockroach, have asthma, and a positive cockroach Nasal Allergen Challenge (NAC) before treatment randomization will be enrolled.

ELIGIBILITY:
Inclusion Criteria:Subject(s)

* And/or parent guardian must be able to understand and provide informed consent;
* Age at date of recruitment (e.g., screening): 8 to 17 years of age
* Have a primary place of residence in one of the pre-selected recruitment census tracts (Reference: Inner-City Asthma Consortium):

  --Note: Subjects who do not live in the pre-selected census tracts but live within the Office of Management and Budget (OMB) defined Metropolitan Statistical Area and have publicly-funded health insurance will qualify for inclusion.
* Have a history of persistent asthma, for a minimum of 1 year before study entry:

  * A diagnosis of asthma will be defined as a report by the caretaker that the subject had a clinical diagnosis of asthma made by a clinician ≥1 year ago, resulting in a prescription of preventative asthma medication, and
  * Must have persistent asthma as defined by the current need for at least 88 mcg fluticasone (or the equivalent of another inhaled corticosteroid) to control asthma at the time of screening.
* At the time of randomization, the subject's asthma must be well controlled as defined by:

  * A Forced Expiratory Volume in 1 second (FEV1) ≥80% predicted, and
  * An Asthma Control Test (ACT) or Childhood Asthma Control Test (CACT) score ≥20.
* Is sensitive to German cockroach as documented by:

  * a positive (≥3 mm greater than negative control) skin prick test result, and
  * detectable German cockroach specific Immunoglobulin E (IgE) (≥ 0.35 kUA/L).
* Have no known contraindications to therapy with glycerinated German cockroach allergenic extract or placebo;
* Have a positive cockroach nasal challenge, as defined by reaching a Total Nasal Symptom Score (TNSS) of ≥6 or a sneezing score of 3 at dose 2 or above during the challenge before randomization; and
* Have documentation of current medical insurance with prescription coverage at randomization.

Exclusion Criteria:Subject(s)

* Unable or unwilling to give written informed consent or comply with the study protocol;
* That is pregnant or lactating;
* That are post-menarcheal females must be abstinent or use a medically acceptable birth control method throughout their participation in the study (e.g. oral, subcutaneous, mechanical, or surgical contraception);
* That cannot perform spirometry and peak flow at treatment randomization;
* That have an asthma severity classification at the time of treatment randomization of severe persistent, using the The National Asthma Education and Prevention Program (NAEPP) classification, as evidenced by at least one of the following:

  * Requires a dose >500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid,
  * Has received more than 2 courses of oral or parenteral corticosteroids in the last 12 months or one course within the last 3 months prior to study entry,
  * Has been treated with depot steroids within the 3 months prior to study entry,
  * Has been hospitalized for asthma within the 6 months prior to study entry, or
  * Has had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to study entry.
* Does not have access to a phone (needed for scheduling appointments);
* Has received allergen immunotherapy (Sublingual Immunotherapy [SLIT] or Subcutaneous Immunotherapy [SCIT]) in the last 12 months or, who plan to initiate or resume allergen immunotherapy during the study;
* Has received biologic therapy (e.g., anti-Immunoglobulin E [IgE], anti-IL-4, anti-IL-5) within 6 months of study entry;
* Has received an investigational drug in the 30 days prior to recruitment or who plan to use an investigational drug during the study;
* Has past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may:

  * pose additional risks from participation in the study,
  * may interfere with the subject's ability to comply with study requirements, or
  * that may impact the quality or interpretation of the data obtained from the study.
* Who have nasal polyps or other major structural abnormalities in their nasal cavities as assessed by anterior rhinoscopy,
* Who meet any of the following criteria are not eligible for enrollment and may not be reassessed:

  * That plan to move from the area during the study period,
  * Have a history of anaphylaxis grade 3 or higher as defined by World Allergy Organization Subcutaneous Immunotherapy Systemic Reaction Grading System,
  * Have unstable angina, significant arrhythmia, uncontrolled hypertension, history of autoimmune disease, or other chronic or immunological diseases that, in the opinion of the investigator, might interfere with the evaluation of the investigational product or pose additional risk to the subject,
  * Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator,

    * may pose additional risks from participation in the study,
    * may interfere with the subject's ability to comply with study requirements,
    * or that may impact the quality or interpretation of the data obtained from the study.
  * Are using tricyclic antidepressants or beta-adrenergic blocker drugs (both oral and topical).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Study Chair — Johns Hopkins Children's Center: Department of Allergy & Immunology; Edward M. Zoratti, MD, Study Chair — Henry Ford Health System: Division of Allergy and Immunology
Locations (11):
- United States (11):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center - IMPACT DC, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System: Division of Allergy and Immunology, Detroit, Michigan
  - St. Louis Children's Hospital: Allergy, Immunology and Pulmonary Medicine Program, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical School, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access will be made available to the public at some point in the future via the mechanism of the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data with the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- [Derived] da Silva Antunes R, Sutherland A, Abawi A, Frazier A, Pomes A, Glesner J, Slater JE, Mindaye ST, Cho K, Zhou G, Ozanne MV, Calatroni A, Visness CM, Altman MC, Wood RA, O'Connor GT, Pongracic JA, Khurana Hershey GK, Kercsmar CM, Gruchalla RS, Gill M, Searing D, Liu AH, Zoratti E, Kattan M, Busse PJ, Sheehan W, Bacharier LB, Teach SJ, Wheatley LM, Togias A, Busse WW, Jackson DJ, Sette A. Cockroach immunotherapy modulates dominant T-cell responses independent of allergen extract content. J Allergy Clin Immunol. 2025 Nov;156(5):1303-1313. doi: 10.1016/j.jaci.2025.07.011. Epub 2025 Jul 24. PMID 40714043
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Inner-City Asthma Consortium — https://www.niaid.nih.gov/clinical-trials/inner-city-asthma-consortium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 308 participants with the goal of enrolling 80 participants into this trial. Each participant received a 12 month treatment.
Groups:
- Cockroach SCIT: Subcutaneous immunotherapy (SCIT): German cockroach allergenic extract. 40 participants 8 to 17 years of age will be randomized to this treatment arm.
  -In the first stage of dose escalation, up to 2 doses of the assigned SCIT treatment will be given weekly, separated by a minimum of 2 days. During the second phase of dose escalation, up to 1 dose of the assigned SCIT treatment will be given weekly, separated by a minimum of 5 days. After maintenance dose is achieved, participants will receive two additional maintenance level-doses spaced approximately 2 weeks apart, followed by maintenance injections every 4 weeks for the remainder of the treatment period. The treatment is for a period of 12 months.
  German cockroach allergenic extract: Active ingredient: a non-standardized allergen derived from the extraction and purification of proteins from German cockroach (Blattella germanica). Non-standardized glycerinated German cockroach allergenic extract is approved in the United States for diagnostic skin testing and immunotherapy by subcutaneous injection (U.S. License 467).
- Placebo: Subcutaneous immunotherapy (SCIT): Placebo for German cockroach allergenic extract. 40 participants 8 to 17 years of age will be randomized to this treatment arm.
  -In the first stage of dose escalation, up to 2 doses of the assigned SCIT treatment will be given weekly, separated by a minimum of 2 days. During the second phase of dose escalation, up to 1 dose of the assigned SCIT treatment will be given weekly, separated by a minimum of 5 days. After maintenance dose is achieved, participants will receive two additional maintenance level-doses spaced approximately 2 weeks apart, followed by maintenance injections every 4 weeks for the remainder of the treatment period. The treatment is for a period of 12 months.
  Placebo for German cockroach allergenic extract: Commercially- labeled licensed product, sterile diluent for allergenic extract (50% glycerinated), sodium bicarbonate (0.091%) sodium chloride (0.166%).
Period: Overall Study
Arm/Group | Cockroach SCIT | Placebo
Started | 40 | 42
Completed | 28 | 29
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 2 | 6
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Moved out of town | 1 | 0
Not completed — >2 bursts of systemic corticosteroids for asthma during treatment period (Starting Nov 2020) | 1 | 2
Not completed — Did not meet randomization criteria | 1 | 1
Not completed — Potential inability to tolerate maintenance dose | 1 | 0
Not completed — Need for dose >500 mcg of fluticasone for 6 months | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population with available data
Groups:
- Total: Total of all reporting groups
Arm/Group | Cockroach SCIT | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (2.48) | 12.2 (2.49) | 12.1 (2.46)
Age, Customized [Count of Participants; unit: Participants]
  Between 8 and 11 years | 12 | 11 | 23
  ≥ 12 years | 16 | 18 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 16 | 37
  White | 2 | 5 | 7
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57
Caretaker completed high school [Count of Participants; unit: Participants] — Measure of Primary Caretaker completed high school
  Participants
    Yes | 23 | 23 | 46
    No | 5 | 6 | 11
Annual household income (<15k) [Count of Participants; unit: Participants] — Category of annual household income that falls below $15,000 per year. Population: Count of participants with an annual household income that falls below $15,000 per year.
  Participants
    Yes | 12 | 16 | 28
    No | 15 | 13 | 28
    Dont Know | 1 | 0 | 1
Cockroach-specific IgE at Baseline [Median (Inter-Quartile Range); unit: kUA/L] — Cockroach-specific IgE Category at Baseline Population: Insufficient blood volume led to missing data for 2 participants.
  kUA/L
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 7.9 [2.4 to 49.2] | 2.6 [0.8 to 12.3] | 4.6 [1.5 to 35.2]
Cockroach-specific IgG4 at Baseline [Median (Inter-Quartile Range); unit: ng/mL] — Cockroach-specific IgG4 at screening Population: Insufficient blood volume led to missing data for 2 participants.
  ng/mL
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 35.0 [35.0 to 207.5] | 35.0 [35.0 to 80.0] | 35.0 [35.0 to 95.0]
NAC responsive dose at baseline [Count of Participants; unit: Participants] — Subjects receive increasing doses of allergens, administered at defined time intervals (every 10-20 minutes) until they react to a dose. A reactive dose is determined when the Total Nasal Symptom Score exceeds 6 or if the subject sneezes 5 or more times. The Total Nasal Symptom Score (TNSS), with a possible score range of 0-12, is the sum of three participant-assessed symptom scores for rhinorrhea, nasal congestion, and nasal itching, as well as a staff-monitored sneezing count. Each symptom is rated on a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe.
  Participants
    Reactive Dose 1 at NAC Baseline - 0 mcg/mL | 0 | 0 | 0
    Reactive Dose 2 at NAC Baseline - 0.00492 mcg/mL | 2 | 2 | 4
    Reactive Dose 3 at NAC Baseline - 0.0155 mcg/mL | 3 | 3 | 6
    Reactive Dose 4 at NAC Baseline - 0.0490 mcg/mL | 1 | 1 | 2
    Reactive Dose 5 at NAC Baseline - 0.155 mcg/mL | 4 | 2 | 6
    Reactive Dose 6 at NAC Baseline - 0.489 mcg/mL | 5 | 6 | 11
    Reactive Dose 7 at NAC Baseline - 1.54 mcg/mL | 6 | 3 | 9
    Reactive Dose 8 at NAC Baseline - 4.88 mcg/mL | 3 | 9 | 12
    Reactive Dose 9 at NAC Baseline - 15.4 mcg/mL | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Total Nasal Symptom Score (TNSS) From Baseline to 12 Months Between Cockroach SCIT and Placebo
Description: The study's primary endpoint is the mean TNSS change from baseline to 12 months, calculated as the difference between baseline and 12-month mean TNSS up to baseline responsive dose. TNSS (0-12) is the sum of three participant-assessed scores for rhinorrhea, congestion, itching, and staff-monitored sneezing, rated 0=None, 1=Mild, 2=Moderate, 3=Severe. Analysis uses ANCOVA modeling mean TNSS difference with factors for treatment arm, site, and baseline mean TNSS. Least square means (LSmeans), SEs, difference in LSmeans between treatment and placebo groups, 95% CI, and p-value are reported. A greater change in the LSmeans indicates a better outcome.
Time Frame: After 12 months
Population: All participants who are randomized, received at least one dose of study treatment, and receive at least one dose during the 12-month NAC.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 28 | 29
score on a scale | -1.02 (0.37) | -0.79 (0.35)
Statistical Analysis 1: Comparison: Cockroach SCIT vs Placebo; Test type: Superiority — The comparison between arms will be conducted using an analysis of covariance (ANCOVA) model, in which the change from the baseline to the 12-month TNSS mean serves as the outcome. The ANCOVA model will incorporate factors for treatment while adjusting for both the baseline TNSS mean and site; p = 0.63, ANCOVA; Least Square Mean Difference = -0.23, 95% CI 2-sided [-1.15 to 0.70]

2. Secondary Outcome: Number of Immunotherapy Related Adverse Events and Number of Immunotherapy Related Serious Adverse Events in the Course of Treatment.
Description: Summary tables will present the total number of Immunotherapy related adverse event within the course of treatment.
Time Frame: After 12 months
Population: All participants who sign consent and undergo study procedures at Screening.
Measure: Number; unit: Adverse Events
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 40 | 42
Adverse Events
  Number of Immunotherapy Related Adverse Events | 130 | 36
  Number of Immunotherapy Related Serious Adverse Events | 0 | 0

3. Secondary Outcome: Change in Area Under the Curve (AUC) Total Nasal Symptom Score (TNSS) From Baseline to 12 Months Between Cockroach SCIT and Placebo
Description: The Total Nasal Symptom Score (TNSS) Area under the curve (AUC) will be calculated separately at baseline and 12 months for each subject using the trapezoidal rule and divided by their baseline reactive dose. TNSS (0-12) is the sum of three participant-assessed scores for rhinorrhea, congestion, itching, and staff-monitored sneezing, rated 0=None, 1=Mild, 2=Moderate, 3=Severe. Analysis uses ANCOVA modeling AUC TNSS with factors for treatment arm, site, and baseline TNSS AUC. Least square means (LSmeans), SEs, difference in LSmeans between treatment and placebo groups, 95% CI, and p-value are reported. A greater change in the LSmeans indicates a better outcome.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 28 | 29
score on a scale | -0.65 (0.33) | -0.48 (0.31)
Statistical Analysis 1: Comparison: Cockroach SCIT vs Placebo; Test type: Superiority; p = 0.69, ANCOVA; Least Square Means Difference = -0.17, 95% CI 2-sided [-0.99 to 0.66]

4. Secondary Outcome: Change in 12-month Responsive Dose Between Cockroach SCIT and Placebo
Description: The 12-month responsive dose is being calculated as the first dose that triggers a reaction of TNSS (Total Nasal Symptom Score) greater than or equal to 6 or a sneeze score of 3, whichever occurs first, in a sequence of up to 9 doses. To estimate the hazard ratio and 95% confidence interval, we are conducting an analysis using Cox regression with censoring, while controlling for the baseline responsive dose and site. Participants who do not experience a reaction before reaching the last dose will be considered right-censored.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 28 | 29
Participants
  Reactive Dose 1 at 12 Months - 0 mcg/mL | 2 | 0
  Reactive Dose 2 at 12 Months -0.00492 mcg/mL | 1 | 0
  Reactive Dose 3 at 12 Months - 0.0155mcg/mL | 1 | 3
  Reactive Dose 4 at 12 Months - 0.0490 mcg/mL | 3 | 1
  Reactive Dose 5 at 12 Months - 0.155 mcg/mL | 1 | 4
  Reactive Dose 6 at 12 Months - 0.489 mcg/mL | 4 | 1
  Reactive Dose 7 at 12 Months - 1.54mcg/mL | 1 | 7
  Reactive Dose 8 at 12 Months - 4.88 mcg/mL | 1 | 3
  Reactive Dose 9 at 12 Months - 15.4 mcg/mL | 14 | 10
Statistical Analysis 1: Comparison: Cockroach SCIT vs Placebo; Test type: Superiority; p = .51, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.42 to 1.54] — At the reactive dose of 15.4 mcg/mL after 12 months, there were 11 participants who were right-censored in the Cockroach SCIT arm and 8 participants who were right-censored in the Placebo arm

5. Secondary Outcome: Change in Log-transformed German Cockroach-specific IgE From Baseline to 12 Months Between Cockroach SCIT and Placebo
Description: The difference in log-transformed German Cockroach-specific IgE between baseline and 12 months is being modeled using ANCOVA with factors for treatment arm, site, and the respective log-transformed IgE baseline as covariates. For each treatment group, we present least square means (LSmeans) and their associated standard errors (SEs). We report the difference in LSmeans between the treatment and placebo groups, along with the associated 95% confidence interval (CI) and p-value.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log(kuA/L)
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 26 | 29
Log(kuA/L) | -0.56 (0.20) | -0.53 (0.19)
Statistical Analysis 1: Comparison: Cockroach SCIT vs Placebo; Test type: Superiority; p = 0.91, ANCOVA; Least Square Means Difference = -0.03, 95% CI 2-sided [-0.54 to 0.49]

6. Secondary Outcome: Change in Log-transformed German Cockroach-specific IgG4 From Baseline to 12 Months Between Cockroach SCIT and Placebo
Description: The difference in log-transformed German Cockroach-specific IgG4 between baseline and 12 months is being modeled using ANCOVA with factors for treatment arm, site, and the respective log-transformed IgG4 baseline as covariates. For each treatment group, we present least square means (LSmeans) and their associated standard errors (SEs). We report the difference in LSmeans between the treatment and placebo groups, along with the associated 95% confidence interval (CI) and p-value.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log(ng/mL)
Arm/Group | Cockroach SCIT | Placebo
Number analyzed (Participants) | 26 | 29
Log(ng/mL) | -1.58 (0.22) | -6.90 (0.21)
Statistical Analysis 1: Comparison: Cockroach SCIT vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least Square Means Difference = 5.32, 95% CI 2-sided [4.77 to 5.87]

7. Other Pre Specified Outcome: EXPLORATORY: Composite Asthma Severity Score (CASI)-by Treatment Group
Description: The Composite Asthma Severity Index (CASI) is a comprehensive severity scale combining multiple facets of asthma severity: impairment, risk, and treatment. The CASI score ranges from 0 to 20 points, with higher scores indicating higher levels of severity, and includes 5 domains: day symptoms and albuterol use, night symptoms and albuterol use, controller treatment, lung function measures, and exacerbations.
Time Frame: Month 10, Month 12
Reporting Status: Not Posted

8. Other Pre Specified Outcome: EXPLORATORY: Number of Days With Asthma Symptoms-by Treatment Group
Description: Defined by the presence of wheezing or tightness in the chest, or cough.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: EXPLORATORY: Number of Nights With Asthma Symptoms-by Treatment Group
Description: Defined by participant waking up during the night due to the presence of wheezing or tightness in the chest, or cough.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: EXPLORATORY: Number of Days With Albuterol Use-by Treatment Group
Description: Albuterol is a bronchodilator used for asthma control.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: EXPLORATORY: Number of Nights With Albuterol use-by Treatment Group
Description: Albuterol is a bronchodilator used for asthma control.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: EXPLORATORY: Asthma Treatment step-by Treatment Group
Description: Defined by medication requirements for asthma control.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: EXPLORATORY: Number of Asthma exacerbations-by Treatment Group
Description: Asthma exacerbation defined as a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the study.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: EXPLORATORY: Spirometry Measurement: Forced Expiratory Volume in 1 Second (FEV1)-by Treatment Group
Description: FEV1 is air volume exhaled in 1 second during spirometry and is a measure of asthma severity.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: EXPLORATORY: Comparison of Rhinitis Symptom severity-by Treatment Group
Description: Measured using the Modified Rhinitis Symptom Utility Index.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: EXPLORATORY: Comparison of Rhinitis Treatment step-by Treatment Group
Description: Defined by medication requirements for rhinitis control.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: EXPLORATORY: Change in German Cockroach-Specific Serum IgG Over Time-by Treatment Group
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin G (IgG) vs. post-baseline German cockroach-specific serum IgG. Numerator is geometric mean post-baseline IgG; denominator is baseline IgG.This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

18. Other Pre Specified Outcome: EXPLORATORY: Change in German Cockroach-Specific Component Allergens Over time-by Treatment Group
Description: Including but not limited to the following component allergens: Bla g 1, Bla g 2, Bla g 4, Bla g 5 and Per a 7.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

19. Other Pre Specified Outcome: EXPLORATORY: Change in Cockroach Skin Test Reactivity Over Time-by Treatment Group
Description: As a measure of response to cockroach immunotherapy.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

20. Other Pre Specified Outcome: EXPLORATORY: Change in Cockroach-Specific Blocking Antibodies Over Time-by Treatment Group
Description: To explore serum measurement(s) of in-vitro cockroach antigen binding to B-cells.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

21. Other Pre Specified Outcome: EXPLORATORY: Change in Cockroach-Specific T Cell Response-by Treatment Group
Description: Limited to Part A only: Peripheral blood mononuclear cells (PBMCs) will be evaluated for the magnitude and phenotype of the Cockroach (CR)-specific T cell response to CR immunotherapy.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

22. Other Pre Specified Outcome: EXPLORATORY: Change in Peripheral Blood Mononuclear Cells (PBMCs) Gene Expression Response to Cockroach (CR) Stimulation Over Time-by Treatment Group
Description: To identify the changes in PBMC gene expression response to cockroach stimulation over time and compare those changes between the treated (German cockroach allergenic extract ) and untreated (placebo) group.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

23. Other Pre Specified Outcome: EXPLORATORY: Change in Nasal Lavage Gene Expression Over Time-by Treatment Group
Description: To identify the changes in nasal lavage gene expression response to cockroach stimulation over time and compare those changes between the treated (German cockroach allergenic extract ) and untreated (placebo) group.
Time Frame: Baseline (Pre-treatment) through Study Completion, an Average of 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (including SAEs) were collected from the time of obtaining informed consent until 30 days after a participant completed study participation or until 30 days after the participant prematurely withdrew or was withdrawn from the study.
Description: The same as clinicaltrials.gov
Arm/Group | Cockroach SCIT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/42
Other Adverse Events (participants affected / at risk) | 34/40 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cockroach SCIT (N=40) | Placebo (N=42)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cockroach SCIT (N=40) | Placebo (N=42)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (3) | 4 (7)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Injection site erythema (General disorders) | 11 (40) | 4 (5)
Injection site haemorrhage (General disorders) | 3 (4) | 0 (0)
Injection site induration (General disorders) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 18 (49) | 3 (3)
Injection site swelling (General disorders) | 4 (5) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 5 (6) | 2 (2)
Food allergy (Immune system disorders) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 5 (7) | 7 (7)
Corona virus infection (Infections and infestations) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 10 (15)
Viral infection (Infections and infestations) | 2 (2) | 5 (5)
Peak expiratory flow rate decreased (Investigations) | 4 (7) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 10 (12) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (8) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03541187/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03541187/SAP_001.pdf